CLINICAL TRIAL: NCT02409264
Title: The Effect of Individualised Homeopathic Treatment of Insomnia Disorder in Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr, University of Johannesburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JessicaLeske201005638
Record Dates: First submitted 2015-03-31; First posted 2015-04-06 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Insomnia Disorder
Keywords: Insomnia; Females; Homeopathy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Individualised Homeopathic Remedy (Experimental): Sucrose pillules will be medicated with the determined individualised homeopathic remedy, in the potency decided by the researcher in accordance with the laws that govern homeopathic prescribing. The dose and repetition of the remedy will be determined by the researcher in accordance with the aforementioned laws. A remedy will be prescribed every 2 weeks, after its determination by the researcher. No remedy will be prescribed after week 8.
  Interventions: Other: Individualised Homeopathic Remedy

INTERVENTIONS:
Other: Individualised Homeopathic Remedy — Sucrose pillules will be medicated with the individualised homeopathic remedy as determined by the researcher, in the potency, dosage and repetition determined by the researcher in accordance with the laws governing homeopathic prescribing.

SUMMARY:
In South Africa, 27% of adult males and 31% of adult females experience insomnia. Insomnia may lead to feelings of fatigue and sleepiness, mood disturbances, cognitive difficulties, and may exacerbate symptomatology of co-morbid diseases. Current conventional treatment for insomnia includes both psychological and drug therapies. These conventional medications potentially may lead to dependency and withdrawal symptoms. Individualised homeopathic treatment is a process in which a homeopath selects the most appropriate remedy for the treatment of a condition in accordance with the fundamental principles of homeopathy. This treatment protocol may offer safe and effective treatment for insomnia disorder, however, more research is required on the subject. The aim of this study is to determine the effect of individualised homeopathic treatment of insomnia disorder in females using detailed case studies and the Insomnia Severity Index.

DETAILED DESCRIPTION:
This study will be of an embedded mixed method case study design, conducted at the University of Johannesburg Doornfontein Homeopathic Health Clinic over a period of 8 weeks. Ten female participants, aged 18 to 45 years, will be recruited by means of non-probability purposive sampling via advertisements placed in the University of Johannesburg Homeopathic Health Clinic and in pharmacies around Johannesburg, with the relevant permission given.

The nature of the study, as well as the requirements for participation will be fully explained and the volunteers will be asked to sign the Participant Information and Consent Form once they agree to participate. Potential participants will undergo a brief screening to determine if they meet the requirements for this study. The participants that meet the inclusion criteria will attend the initial consultation and those that do not meet the inclusion criteria will be referred to the Homeopathic Health Clinic.

The consultation will consist of a comprehensive homeopathic case history, the conduction of relevant physical exams, including vital signs, and the completion of the Insomnia Severity Index (ISI). The participant's case will be analysed and computer repertorised, using the Complete Repertory of Mercurius homeopathic software (Aeon Group), version 5.3.0.17. The individualised homeopathic remedy will be selected by the researcher who will refer to the appropriate Materia Medica. The Homeopathic Dispenser will dispense the homeopathic remedy to the participant.

Each participant will return for four follow-up consultations which will be two weeks apart. At each follow-up consultation the ISI will be completed and a follow-up case history and physical examination of the participants' vital signs will be conducted. The participants' symptoms will be re-evaluated and a remedy prescribed accordingly. At the final consultation in the 8th week, no remedy will be prescribed.

Data will be collected and analysed by the researcher with the assistance of a statistician at Statkon, using non-parametric tests, including: frequencies and descriptives, the Friedman test, and Wilcoxon post hoc test.

The possible outcome of this study may demonstrate that individualised homeopathic treatment is effective in reducing the frequency and intensity of insomnia disorder in females, and instigate further research on the subject.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years to 45 years.
* Participants must fulfil the diagnostic criteria for insomnia disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition Text Revision (DSM-V TR):

  * A predominant complaint of dissatisfaction with sleep quantity or quality, associated with one (or more) of the following symptoms: difficulty initiating sleep; difficulty maintaining sleep, characterized by frequent awakenings or problems returning to sleep after awakenings; and/or early-morning awakening with inability to return to sleep
  * The sleep disturbance causes clinically significant distress or impairment in social, occupational, educational, academic, behavioural, or other important areas of functioning
  * The sleep difficulty occurs at least 3 nights per week
  * The sleep difficulty is present for at least 3 months
  * The sleep difficulty occurs despite adequate opportunity for sleep
  * The insomnia is not better explained by and does not occur exclusively during the course of another sleep-wake disorder (e.g., narcolepsy, a breathing-related sleep disorder, a circadian rhythm sleep-wake disorder, a parasomnia)
  * The insomnia is not attributable to the physiological effects of a substance (e.g., a drug of abuse, a medication)
  * Coexisting mental disorders and medical conditions do not adequately explain the predominant complaint of insomnia.

Exclusion Criteria:

* Pregnant or lactating women
* Participants suffering from narcolepsy, a breathing-related sleep disorder, circadian rhythm sleep disorder, or a parasomnia
* Participants diagnosed with major depressive disorder, generalised anxiety disorder, a delirium, or schizophrenia
* Participants using conventional psychological or drug therapies, or herbal, or homeopathic medication for their insomnia
* Participants taking recreational or prescription drugs which have insomnia as a side effect.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Every 2 weeks for 8 weeks
  The Insomnia Severity Index is a 7-item questionnaire that provides a global measure of an individual's perceived insomnia severity.

SECONDARY OUTCOMES:
Qualitative case history notes | Every 2 weeks for 8 weeks
  Case notes taken by the researcher with regard to the participants' symptoms, characteristics and wellbeing, which are used to determine the individualised homeopathic remedy and collect qualitative data from each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Pellow, M.TechHom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa